CLINICAL TRIAL: NCT06844695
Title: The Effects of Virtual Museum Visit With Virtual Reality Glasses on Pain, Fatigue, and Anxiety in Patients Receiving Chemotherapy: A Randomized Controlled Trial
Brief Title: Effects of Virtual Museum Visit on Pain, Fatigue, and Anxiety in Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Mukadder Mollaoğlu, Prof. Dr., Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SCUniv
Record Dates: First submitted 2025-02-14; First posted 2025-02-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy Effect; Pain Cancer; Fatigue; Anxiety
MeSH Terms: conditions — Cancer Pain; Fatigue; Anxiety Disorders | interventions — Art Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Art Therapy Intervention Group (Experimental): The Intervention Group is informed about how to use the virtual glasses and is tested. One week after the first test, the patients in the Intervention Group visit a virtual museum on the theme of the patients' choice for an average of 20 minutes using virtual glasses for a total of five consecutive weeks. In the fifth virtual tour session, which is the third and final application session, measurements (Visual Analog Scale, Hirai Cancer Fatigue Scale and Beck Anxiety Scale) are made in both groups.
  Interventions: Other: Art Therapy (Virtual Museum Visit)
- No Intervention: Control Group (No Intervention): No virtual museum visit was applied to the control group. Scales were applied to individuals. For the control group, evaluations were made with scales three times in total.

INTERVENTIONS:
Other: Art Therapy (Virtual Museum Visit) — Virtual Reality (VR) is a technology that creates simulated settings in which users can interact and experience as if they were physically there.Virtual Reality typically involves the use of a headset or glasses that display the virtual environment, as well as other input devices such as controllers or gloves that allow users to interact with the virtual world
  Arms: Experimental: Art Therapy Intervention Group

SUMMARY:
Symptom management is the most important aspect of clinical cancer care. Virtual reality-based interventions can be used to improve cancer patients' experiences with medical treatment, with their distraction-based effects. The aim of this study was to determine the effects of virtual museum visits with virtual reality glasses on pain, fatigue, and anxiety in patients receiving chemotherapy. The study included a museum visit with virtual reality glasses during the procedure in addition to routine treatments for patients in the intervention group. Patients in the control group were given only their routine treatments. Data will be collected using the Personal Information Form (PIF), Hirai Cancer Fatigue Scale, Visual Analog Scale (VAS) and Beck Anxiety Scale (BAÖ). In the first interview, the patient was also presented with virtual museum options and the museums he/she wanted to visit were listed. In addition, the patients in the Intervention Group were shown virtual museums with 53 different themes on the website prepared by the General Directorate of Information Technologies of the Ministry of Culture and Tourism, which is located on the website ''https://sanalmuze.gov.tr'' belonging to the Ministry of Culture and Tourism, and the museums they wanted to visit in each session according to their preferences were listed. In the meantime, the Intervention Group was explained how to use the virtual glasses and they will be tested. One week after the first test, the patients in the Intervention Group will visit a virtual museum on the theme preferred by the patients using virtual glasses for an average of 20 minutes for a total of five consecutive weeks. In the fifth virtual tour session, which is the third and last application session, measurements (Visual Analog Scale, Hirai Cancer Fatigue Scale and Beck Anxiety Scale) will be administered. The control group will not receive any intervention other than routine treatment.The museum visit applied to the Intervention Group will also be applied to the control group after the study is completed, taking into account the ethical dimension.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of the sample were having received at least one course of chemotherapy and continuing chemotherapy
* Having not visited a virtual museum with VR glasses before,
* Having no difficulty in communicating,
* Having no mental problems, being 18 years of age or older,
* Agreeing to participate in the study

Exclusion Criteria:

* The exclusion criteria of the sample were having not received chemotherapy or having completed treatment.
* Having Stage IV cancer
* Having difficulty seeing and communicating.
* Being under the age of 18
* The desire to withdraw from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Hirai Cancer Fatigue Scale | It will take 5 weeks to collect data three times after randomization is done. The first measurement of fatigue scale will be done in the first week, the second measurement in the third week and the third measurement in the fifth week of virtual muse
  The scale, originally named "Hirai Cancer Fatigue Scale", was developed by Kazue Hirai et al. in 2015 and consisted of 15 items . The scale is used to measure fatigue in cancer patients and has a 5-point Likert design. Each item on the scale is evaluated as 1 "not at all", 2 "very little", 3 "a little", 4 "a lot", and 5 "very much". It has 3 sub-dimensions (Physical-Mental, Activity-Related Sensitivity, and Cognitive Sensitivity). Items 1-6 on the scale constitute the Physical-Mental Sub-Dimension, items 7-12 constitute the Activity-Related Sensitivity Sub-Dimension, and items 12-15 constitute the Cognitive Sensitivity Sub-Dimension. The scale has no cut-off point. The minimum value of the scale is 15 and the maximum value is 75, with high scores indicating increased fatigue, while low scores indicating less fatigue. The validity and reliability study in our country was conducted by Mencel.
Visual Analog Scale (VAS) | It will take 5 weeks to collect data three times after randomization is done. The first measurement of VAS will be done in the first week, the second measurement in the third week and the third measurement in the fifth week of virtual museum visit.
  VAS, which evaluates the intensity of pain, is widely used in adults. The scale was developed by Price et al. as a scale consisting of a single 10 mm line that evaluates the intensity of pain. The two end definitions of the parameter to be evaluated are written at both ends of the line and the patient is asked to indicate where his/her condition is appropriate on this line by drawing a line, putting a dot, or pointing. For example, for pain, no pain is written at one end and very severe pain is written at the other end and the patient marks his/her current condition on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain. It has been shown that the line on which the test is applied is not affected by whether it is horizontal or vertical or by its length. The average of the values obtained for the patients is taken.
Beck Anxiety Inventory (BAI) | It will take 5 weeks to collect data three times after randomization is done. The first measurement of BAI will be done in the first week, the second measurement in the third week and the third measurement in the fifth week of virtual museum visit.
  The inventory was developed by Beck et al. to determine the level and frequency of anxiety symptoms experienced by individuals. The scale has a Likert design with self-assessment consisting of 21 items and is scored between 0-3. The high total score indicates the high level of anxiety experienced by the individual. The score range varies between 0-63. The scale is evaluated as 0-7 points, no anxiety symptoms, 8-15 points, mild anxiety, 16-25 points, moderate anxiety, 26-63 points, and severe anxiety symptoms. The validity and reliability study in our country was conducted by Ulusoy et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Mukadder, Mollaoğlu, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 25 May 2025

REFERENCES:
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Hirai K, Kanda K, Takagai J, Hosokawa M. Development of the Hirai Cancer Fatigue Scale: Testing its reliability and validity. Eur J Oncol Nurs. 2015 Aug;19(4):427-32. doi: 10.1016/j.ejon.2014.12.004. Epub 2015 Feb 2. PMID 25656217
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917